CLINICAL TRIAL: NCT01726088
Title: A Double-Blind, Placebo-Controlled Trial of Modafinil in OEF/OIF Combat Veterans With PTSD
Brief Title: Modafinil in the Treatment of PTSD (Posttraumatic Stress Disorder)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biomedical Research Foundation (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Timothy Kimbrell, Staff Physician; Associate Professor, Biomedical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAVHS209470-1; 5P20RR020146-09 (NIH); 8P20GM103425-09 (NIH)
Record Dates: First submitted 2012-08-03; First posted 2012-11-14 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Modafinil; p50; Attentional Bias
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- modafinil (Active Comparator): Study participants randomized to the active arm of the study will take modafinil 100mg capsules orally each day for 4 weeks.
  Interventions: Drug: Modafinil
- Sugar Pill (Placebo Comparator): Study participants randomized to the placebo arm of the study will take matching capsules orally each day for 4 weeks.
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: Modafinil — we will compare the effect of modafinil and matching placebo on clinical and objective measures detailed above.
  Other Names: Provigil

SUMMARY:
The purpose of this study is to determine if modafinil is more effective than placebo in the treatment of posttraumatic stress disorder (PTSD) in male combat veterans who have been deployed to Iraq or Afghanistan.

DETAILED DESCRIPTION:
There is a high rate of posttraumatic stress disorder (PTSD) in soldiers exposed to combat in Operations Enduring Freedom and Iraqi Freedom (OEF/OIF). Unfortunately, currently available treatments for combat-related PTSD have produced modest treatment gains at best. New treatment strategies that can be directed toward objectively measured correlates of PTSD are urgently needed.

Specific Aims: 1) To determine if there is evidence for the effectiveness and tolerability of adjunctive modafinil in the treatment of combat-related PTSD. We hypothesize that OEF/OIF veterans with PTSD randomized to modafinil 100mg/day for four weeks will experience more improvement in PTSD symptoms than OEF/OIF veterans with PTSD randomized to placebo treatment for four weeks. 2) To determine if PTSD symptom severity is associated with electrophysiological and neuropsychological measures of pre-attention and attention and if these measures change to a greater degree in participants randomized to modafinil versus those randomized to placebo. We hypothesize modafinil treatment will result in greater changes in electrophysiological and neuropsychological measures of pre-attention and attention than placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF Veteran with a history of deploying to Afghanistan or Iraq
* right-handed
* male 20-60 years of age
* meets Diagnostic and Statistical Manual (DSM-IV) diagnostic criteria for PTSD
* competent to give informed consent
* access to a telephone
* stable psychotropic medication regimen for a minimum of four weeks prior to enrollment
* able and willing to complete the required schedule of evaluations (Baseline in person, 1 week by phone, 2 week in person, 4 week in person)

Exclusion Criteria:

* diagnosis of schizophrenia, schizoaffective disorder or bipolar disorder
* current substance abuse or dependence
* history of seizure disorder or severe traumatic brain injury
* history of attempted suicide within the previous two years or active suicidal ideation within the past month
* currently taking benzodiazepines except for bedtime dosing only
* currently taking stimulant medication
* known allergic reaction to modafinil or currently taking medication
* that may have altered metabolism if taken with modafinil: Tricyclic antidepressants (amitriptyline; nortriptyline; desipramine; imipramine; CNS stimulants (amphetamine; d-ampthetamine; atomoxetine); Carbamazepine; Phenytoin; Phenobarbitol; Rifampin; Ketaconazole; MAO Inhibitors (isoniazid; selegiline); Warfarin; Diazepam; Mephenytoin; Cyclosporine; Theophylline

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | Change in CAPS from baseline to 4 weeks
  The CAPS is the gold standard measure of PTSD symptoms

SECONDARY OUTCOMES:
eye-gaze tracking to facial stimuli | change in eye-gaze tracking from baseline to 4 weeks
  a measure of attentional bias
Modified Stroop | Change in Modified Stroop from baseline to 4 weeks
  a measure of attentional bias
event related potentials | Change in P50 from baseline to 4 weeks
  P50 potential a measure of level of arousal or pre-attentional processing at 3 interstimulus intervals-ISIs

CONTACTS AND LOCATIONS:
Overall Officials: Tim A Kimbrell, MD, Principal Investigator — Central Arkansas VA Healthcare System
Locations (1):
- CAVHS Eugene Towbin VA Medical Center, North Little Rock, Arkansas, United States